CLINICAL TRIAL: NCT01707654
Title: Repair of Infective Wound Associated With Nerve Defect in the Finger Using A Bipedicled Nerve Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSChen6017; HEBEI-J06451 (Other: Hebei Ethics Committee)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2012-04

CONDITIONS: Infection Wound; Disruption of Nerve Repair
Keywords: defect;; dorsal branch of the proper digital nerve;; proper digital nerve;; finger sensory reconstruction.
MeSH Terms: conditions — Wound Infection

ARMS (1):
- nerve graft (Other): Simultaneous repair of the infected wound and digital nerve defect in the finger using a bipedicled nerve flap including nerve graft from the dorsal branch of the digital nerve.
  Interventions: Device: Nerve flap

INTERVENTIONS:
Device: Nerve flap — Based on the Teoh et al.'s technique, we combined the nerve graft into the bipedicled heterodigital arterialized island flap and used this composite flap tissue for reconstructing complicated infected wound in the finger.

SUMMARY:
A combination of soft tissue and digital nerve defects in the finger results in sensory loss of the finger pulp. Reconstruction of these combined injuries is difficult. When the neurocutaneous defect is associated with wound infection, reconstructive alternatives are more limited. From July 2008 to May 2010, a retrospective study was conducted with 9 consecutive postinfection patients who had the neurocutaneous defect of the finger following trauma. The purpose of this retrospective study is to report repair of the complicated infected wound in the finger using the bipedicled nerve flap and to evaluate the efficacy of this technique.

DETAILED DESCRIPTION:
sensation of the flaps is assessed using static two-point discrimination (2PD) and Semmes-Weinstein monofilament (SWM) testing at final follow-up. The cold intolerance of the injured finger is measured using the self-administered Cold Intolerance Severity Score questionnaire that was rated into mild, moderate, severe, and extreme (0-25, 26-50, 51-75 and 76-100). Patients report their satisfaction with functional recovery of the injured finger according to the Michigan Hand Outcomes Questionnaire that was based on a 5-point response scale.

ELIGIBILITY:
Inclusion Criteria:

* an infective wound with exposed bone or tendon in the finger;
* soft tissue defect involving proximal half of the middle phalanx, the proximal phalanx, or both;
* associated digital nerve defect 1 to 4 cm in length;
* single or double nerve defects; and
* simultaneous repair of nerve and soft tissue defects.

Exclusion Criteria:

* injury to the course of the pedicle or the donor site;
* nerve defect less than 1 cm or larger than 4 cm in length;
* occurrence of the defect in a region the flap is unable to reach, such as distal interphalangeal joint region, distal portion of the middle phalanx of the middle finger and the thumb;
* no involvement of the digital nerve.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Zhang X, Shao X, Gao S, Wang B, Liu D. Treatment of a combination of volar soft tissue and proper digital nerve defects using the dorsal digital nerve island flap. J Hand Surg Am. 2010 Oct;35(10):1655-1662.e3. doi: 10.1016/j.jhsa.2010.07.011. PMID 20888502
- [Derived] Chen C, Tang P, Zhang L. Use of a bipedicled nerve flap taken from the dorsum of the digit for reconstruction of neurocutaneous defect in the adjacent finger. J Plast Reconstr Aesthet Surg. 2013 Oct;66(10):1322-9. doi: 10.1016/j.bjps.2013.06.001. Epub 2013 Jul 2. PMID 23829956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2008 to May 2010, 9 patients who had a combination of soft tissue and digital nerve defects were included in the study. The type of location was medical clinic.
Pre-assignment Details: No patient was lost to follow-up
Period: Overall Study
Arm/Group | Nerve Graft
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nerve Graft
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  China | 9

OUTCOME MEASURES:

1. Primary Outcome: 2-point Discrimination Test
Description: The 2-point Discrimination Test determines the minimal distance at which a subject can sense the presence of two needles. The modified American Society for Surgery of the Hand guidelines were used to stratify Discriminator measurements (excellent <6 mm; good 6-10 mm; fair 11-15 mm; poor >15 mm. The test points were at the center of the radial or ulnar portion of the pulp. Each area was tested 3 times with a Discriminator (Ali Med, Dedham, MA). Two out of 3 correct answers were considered proof of perception before proceeding to another lower value. We stopped at 4 mm as a limit of 2PD and considered this normal. The assessments were performed at a single time point at the final follow up.
Time Frame: 17-25 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Nerve Graft
Number analyzed (Participants) | 9
mm | 7.5 (1.6)

2. Secondary Outcome: Semmes-Weinstein (SW) Monofilament Test
Description: The test points were at the center of the radial or ulnar portion of the pulp. The donor site, i.e. radial- or ulnar-dorsal aspect of the middle phalanx of the donor digit, was also evaluated.
Time Frame: 17-25 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Pain
Description: Pain was given subjectively by the patient using the visual analogue scale (VAS). The VAS consists of a 10 cm line that was grouped into mild (1-3 cm), moderate (4-6 cm) and severe (7-10 cm).
Time Frame: 17-25 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Nerve Graft
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes